CLINICAL TRIAL: NCT03018912
Title: Validating the Use of a Novel Subjectively Reported Sleep Vital Sign for the Identification and Management of Sleep Disorders
Brief Title: Validating the Use of a Subjectively Reported Sleep Vital Sign
Acronym: SSVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Dennis Hwang, MD, Department Medical Director, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: KPSleep-002
Record Dates: First submitted 2016-11-01; First posted 2017-01-12 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea (OSA); Insomnia; Restless Leg Syndrome (RLS); Hypersomnia Type; Sleep Disorder; Shift Work Sleep Disorders
Keywords: Subjective Sleep Vital Sign (VS); Primary Care; Sleep Medicine; Cognitive Behavioral Therapy (CBT); Obstructive Sleep Apnea (OSA); Insomnia; Complex Sleep Disorders; Predictive Analytics; Screening; Therapy Outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders; Restless Legs Syndrome; Disorders of Excessive Somnolence; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep VS (Experimental): Patients check-in for their primary care physician visit and are provided a Sleep VS survey packet. Investigators or research associates will review the Sleep VS, and patients that screen positive on their Sleep VS will be asked to complete an extended set of sleep questions. A triaging algorithm will be available based on answers to the extended sleep questions to assist the primary care physician with assessment and triaging care. Patients that screen "negative" will not be asked the extended sleep questions nor will they be brought to the attention of the primary care physician and proceed with "usual care."
  Interventions: Other: Sleep VS
- Usual Care (No Intervention): Patients check-in for their primary care physician visit and proceed with "usual care". Although the sleep vital sign will not be collected, the medical providers can still use the extended sleep questionnaire and triaging algorithm, if in the course of caring of the patient a potential sleep disorder is recognized.

INTERVENTIONS:
Other: Sleep VS — During check in patients are instructed to complete the Sleep VS survey packet only. The Sleep VS survey packet will take approximately 4 minutes to complete. The packet includes the subjective Sleep VS and additional sleep questionnaires, such as ESS, FOSQ-10, ISI, and sleep-wake pattern questions.
  The subjective Sleep VS is composed of the following 2 questions:
  1. How many days a week are you satisfied with your sleep?
  2. How many days a week is sleepiness a problem?
  Arms: Sleep VS

SUMMARY:
Sleep disorders are commonly under-recognized in the primary care setting and available screening tools are often are limited. The study inestigators hypothesize that the use of a novel subjective sleep vital sign (VS) will improve recognition of patients with sleep disorders and can be utilized to track outcomes to sleep therapy.

DETAILED DESCRIPTION:
Background

The ability to identify patients with sleep disorders is recognized as increasingly important given its association with cardiovascular disease and impact on daytime functioning and quality of life. The Center for Disease Control recently characterized insufficient sleep as a public health issue, while also estimating that 1 in 25 adults admit to falling asleep while driving in a given month. 50 to 70 million Americans are affected by chronic sleep disorders and intermittent sleep problems, yet sleep problems are under-recognized; for example, 80 to 90% of adults with sleep disordered breathing remain undiagnosed. Sleep disorder screening tools are available, but are often limited by the following factors:

1. Surveys may be extensive and thereby limit utilization
2. Screening tools are often targeted for specific sleep disorders (e.g. obstructive sleep apnea (OSA)) rather than to more comprehensively screen for a wide range of sleep disorders
3. Screening tools may not be useful in assessing outcomes during follow-up care

We propose the development of a sleep vital sign (VS) constructed as a simple-to-use survey tool that can assist primary care in identifying patients with sleep disorders and potentially useful to assess response to treatment. Improved identification of sleep disorders can potentially result in a benefit to the individual patient, to the health system, and to the greater public health.

Study Proposal We plan to investigate the use of a sleep VS (subjective patient reported metric) as a potential tool to identify patients with sleep disorders and to measure outcomes during follow-up care.

This pilot study is structured as a 2-arm randomized, prospective clinical trial with the following specific aims:

1. To determine whether subjective sleep vital signs can improve the rate of identifying patients with sleep disorders in a primary care setting.
2. To determine if subjective sleep vital signs can track patient therapy response for various sleep disorders.
3. To correlate subjective sleep vital sign results with validated sleep measurements (e.g. sleep surveys, Continuous Positive Airway (CPAP) usage)

Methods

This study is a 2-arm randomized clinical trial. Patients checking into Kaiser Fontana Medical Center primary care clinics (Internal Medicine), will be randomized into one of the following pathways: Sleep Vital Sign (VS) Pathway or Usual Care (refer to Workflow Figure). We intend to use the first day of recruitment to identify challenges with protocol implementation in a primary care clinic. Data collected during this day will only be used to compare sleep VS to the other validated sleep questionnaires in the survey packet; however, this data will not be used to compare rates of identifying sleep disorders between sleep VS and usual care pathways.

Sleep VS Pathway When enrolling, we plan to inform the patients that we are performing a study pertaining generally to overall well-being and quality of life, while withholding information that the study pertains specifically to screening for sleep disorders. We believe it is necessary to withhold information (incomplete disclosure) that the study is specifically about sleep disorders in order to limit the risk of selection bias. If "sleep disorders" was provided as full disclosure as the topic of the study, it may incentivize patients with sleep problems to participate in the study (while dis-incentivizing those without sleep problems from participating), thus introducing a potential selection bias. Selection bias could affect the determined accuracy of the sleep VS in identifying sleep disorders which is the primary aim of this study, and negatively affect the scientific and educational value of this study. Furthermore, it would limit our understanding on proper practical implementation into healthcare delivery workflows.

At check-in, a research associate will ask patients if they are interested in participating in a research study. If patient expresses interest, the research associate will explain the study and give an informational sheet utilizing an anticipated IRB approved script. Those who have given verbal consent, after reviewing the information sheet, will be provided a Sleep VS survey packet (packet includes: Sleep VS, sleep-wake assessment, ESS, FOSQ-10, and ISI).

Debriefing process: immediately after the patient completes this "Sleep VS survey packet", the investigator will inform the patient that the purpose of this study specifically pertains to discovering tools that may help medical providers better identify patients with sleep disorders and will provide patient with contact for Dr. Dennis Hwang, the study's primary investigator, in the event that the patient wishes to withdraw their data from inclusion in study analysis.

The proposed Sleep VS is based on the following 2 questions:

1. How many days a week are you not satisfied with your sleep?
2. How many days a week is sleepiness a problem?

For the purposes of this study, the Sleep VS will be considered a positive screen if patients response to 1) or 2) is ≥4 days. Investigators or research associates will review the Sleep VS, and patients that screen positive will be:

1. Asked an extended set of sleep questions (refer to Triaging Algorithm Figure)
2. Brought to the attention of the primary care physician.

A triaging algorithm will be available based on answers to the extended sleep questions to assist the primary care physician with assessment and triaging care (refer to Triaging Algorithm Figure). Patients will primarily be triaged to sleep medicine (for OSA assessment, complex insomnia patients, and other patients with more complex sleep disorders), to health education 4-week cognitive behavioral therapy (CBT) program for less complex insomnia or remain under the care of the primary care physician. If the patient is referred to sleep medicine, the sleep VS will be performed at each sleep center appointment (it is already part of our standard usual clinical care). The triaging algorithm is a tool to assist the primary care physician with management suggestions, but the physician has the flexibility to manage the patient according to best clinical judgment.

Patients that screen "negative" will not be asked the extended sleep questions nor will they be brought to the attention of the primary care physician. They will proceed with "usual care." If during the course of "usual care", a potential sleep disorder is discussed, the extended sleep questions with triaging algorithm can still be utilized to assist in determining management.

Usual Care Pathway Patients will not be provided the sleep VS packet during check-in. If during the course of usual care, a potential sleep disorder is discussed, the extended sleep questions with triaging algorithm can still be utilized to assist in determining management at the discretion of the primary care physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have a scheduled office visit with their primary care physician.
* Patients have to be Kaiser Permanente members

Exclusion Criteria:

* Non-English speaking patients unable to understand English to complete the surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Disorder Identification Rates | 3 months
  Compare the rate of identification of sleep disorders between each pathway

SECONDARY OUTCOMES:
Referral Rates | 3 months
  Compare the rate of referrals to sleep medicine, health education, and/or other departments for sleep disorders between each pathway
Sleep VS vs Sleep Questionnaires | Every time patient completes the Sleep VS survey packet over a 3 month period.
  Compare the Sleep VS results with the other establish sleep questionnaires (ESS, FOSQ-10, and ISI) between the Active and Non-Active pathways
Assessing response to treatment using Sleep VS | Every time patient completes the Sleep VS survey packet over a 3 month period.
  Compare Sleep VS at baseline and during follow-up care between the Active and Non-Active pathways, and correlating such assessments with sleep diagnosis and therapy provided.
Medications and Encounters | 3 months
  Compare the use of sleep/psychiatric medications and healthcare encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Sleep Center; Fontana Medical Center, Kaiser Permanente, Fontana, California, United States

IPD SHARING:
Plan to Share IPD: No
This study will be conducted solely within Kaiser Permanente, and it is unnecessary to release IPD to external sources or organizations.

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Sleep Medicine and Research; Colten HR, Altevogt BM, editors. Sleep Disorders and Sleep Deprivation: An Unmet Public Health Problem. Washington (DC): National Academies Press (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK19960/ PMID 20669438